CLINICAL TRIAL: NCT00402857
Title: Advanced Parenting Education in Pediatrics: The APEP Project
Brief Title: Parent Training to Promote Early Identification and Treatment of Childhood Behavioral Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH076244 (NIH); R01MH076244 (NIH); DSIR CT-C
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Attention Deficit and Disruptive Behavior Disorders
Keywords: Parenting Education; Child, Preschool; Preventive Intervention; Primary Health Care; Pediatrics; Attention Deficit Disorders; Oppositional Defiant Disorder; Disruptive Behavior Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Attention Deficit and Disruptive Behavior Disorders; Oppositional Defiant Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive the Incredible Years Program, a group parenting intervention
  Interventions: Behavioral: Incredible Years Program
- 2 (Other): Participants assigned to the waitlist condition will receive the Incredible Years Program after a 1-year waiting period
  Interventions: Behavioral: Incredible Years Program

INTERVENTIONS:
Behavioral: Incredible Years Program — The Incredible Years Program is a 10-week group parenting intervention. Parent training sessions will take place once per week for 10 weeks, and will last approximately 2 hours each. Sessions will focus on teaching positive parenting skills, such as appropriate play and use of praise and rewards, as well as limit-setting techniques, such as ignoring, allowing children to experience the natural consequences of their actions, and assigning time-outs.

SUMMARY:
This study will evaluate the effectiveness of a parent training program in improving parenting skills and reducing behavioral symptoms in young children who are at risk for developing childhood behavior disorders.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) and oppositional defiant disorder (ODD) are common childhood behavior disorders. Children with ADHD experience hyperactivity, distractibility, poor concentration, and impulsivity. If left untreated, ADHD can continue into adulthood, and can cause problems in family, social, and work environments. Children with ODD exhibit an ongoing pattern of uncooperative, defiant, and hostile behavior toward authority figures. Symptoms of ODD, including frequent temper tantrums, anger, resentment, and vindictiveness, may interfere with a child's everyday functioning. The Incredible Years parent training program has been shown to be effective in multiple settings at training parents to manage their child's behavior. This study will evaluate the effectiveness of the Incredible Years training program within a pediatric office setting at improving parenting skills and reducing behavioral symptoms in young children who are at risk for developing childhood behavior disorders.

Participants in this open-label study will be randomly assigned to the Incredible Years training program or a waitlist condition, in which they will begin the program after a 1-year waiting period. Parent training sessions will take place once per week for 10 weeks, and will last approximately 2 hours each. Sessions will focus on teaching positive parenting skills, such as appropriate play and use of praise and rewards, as well as limit-setting techniques, such as ignoring, allowing children to experience the natural consequences of their actions, and assigning time-outs. Self-report assessments and phone interviews will be used to assess outcomes. Additionally, follow-up visits will occur immediately post-intervention and 6 and 12 months post-intervention. Children will attend one visit before the program begins, as well as the follow-ups held immediately post-intervention and 12 months post-intervention. These visits will include videotaped observations of children and their primary caregivers.

ELIGIBILITY:
Inclusion Criteria:

Parent or primary caregiver of a child who fits the following criteria:

* Receives a positive result on behavioral screening

Exclusion Criteria:

Parent or primary caregiver of a child who fits the following criteria:

* Diagnosis of pervasive developmental disorder or global developmental delay

Ages: 22 Months to 38 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 345 (Actual)
Dates: Start 2006-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Parenting behavior | Measured post-intervention and at 6- and 12-month follow-ups
Child disruptive behaviors | Measured post-intervention and at 6- and 12-month follow-ups

SECONDARY OUTCOMES:
Child and parent functional status/impairment | Measured post-intervention and at 6- and 12-month follow-ups
Parenting stress | Measured post-intervention and at 6- and 12-month follow-ups
Family functioning | Measured post-intervention and at 6- and 12-month follow-ups
Consumer perspectives | Measured post-intervention and at 6- and 12-month follow-ups
Cost of services | Measured post-intervention and at 6- and 12-month follow-ups
Barriers to treatment | Measured post-intervention and at 6- and 12-month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Ellen C. Perrin, MD, Principal Investigator — Tufts Medical Center; Christopher Sheldrick, PhD, Principal Investigator — Tufts Medical Center; Jannette McMenamy, PhD, Principal Investigator — Fitchburg State College
Locations (9):
- United States (9):
  - MGH Chelsea Healthcare Center, Chelsea, Massachusetts
  - Codman Square Health Center, Dorchester, Massachusetts
  - Martha Eliot Health Center, Jamaica Plain, Massachusetts
  - Medical Associates Pediatrics, Leominster, Massachusetts
  - Southboro Medical Group, Southborough, Massachusetts
  - Pediatrics West, Westford, Massachusetts
  - Westwood-Mansfield Pediatric Associates, Westwood, Massachusetts
  - Wilmington Pediatrics, Wilmington, Massachusetts
  - Woburn Pediatric Associates, Woburn, Massachusetts

REFERENCES:
- [Derived] Perrin EC, Sheldrick RC, McMenamy JM, Henson BS, Carter AS. Improving parenting skills for families of young children in pediatric settings: a randomized clinical trial. JAMA Pediatr. 2014 Jan;168(1):16-24. doi: 10.1001/jamapediatrics.2013.2919. PMID 24190691